CLINICAL TRIAL: NCT04595266
Title: Randomized, Multicenter Phase II Study of Monoclonal FOLFOX6m + mAb Alone or in Combination With Liver Chemoembolization (Lifepearls-Irinotecan) in Patients With Colorectal Cancer and Metastatic Disease Limited to the Liver With Poor Prognosis
Brief Title: Chemoembolization (Lifepearls-Irinotecan) in Patients With Colorectal Cancer and Metastatic Disease
Acronym: LIVERPEARL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol Multidisciplinario del Cancer Digestivo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEMCAD-1802; 2020-003795-40 (EudraCT Number)
Record Dates: First submitted 2020-10-06; First posted 2020-10-20 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Cancer Metastatic; Liver Metastasis Colon Cancer
Keywords: Colorectal cancer; Chemoembolization; LIVERPEARLS-Irinotecan; Liver metastasis
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol; Leucovorin; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1: 1 ratio in the 2 arms:
  Control Arm. Systemic chemotherapy with FOLFOX6m + monoclonal Ab Experimental Arm. Systemic chemotherapy with FOLFOX6m + monoclonal Ab + Intra-arterial liver chemotherapy with LIFEPEARLS-IRINOTECAN (catheterization and infusion of 100 +/- 50 micron microspheres loaded with 100 mg of irinotecan in both liver lobes) cycles 2 and 4.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Systemic chemotherapy with FOLFOX6m + monoclonal Ab (anti-EGFR or bevacizumab).
  Interventions: Drug: FOLFOX regimen; Biological: Anti-EGFR or Bevacizumab
- Experimental (Experimental): Systemic chemotherapy with FOLFOX6m + monoclonal Ab (anti-EGFR or bevacizumab) + Intra-arterial liver chemotherapy with LIFEPEARLS-IRINOTECAN (catheterization and infusion of 100 +/- 50 micron microspheres loaded with 100 mg of irinotecan in both liver lobes) cycles 2 and 4.
  Interventions: Drug: FOLFOX regimen; Biological: Anti-EGFR or Bevacizumab; Drug: LIVERPEARLS-Irinotecan

INTERVENTIONS:
Drug: FOLFOX regimen — Leucovorin: 400 mg / m2 IV over 15 minutes on day 1 of each cycle. Fluorouracil (5-FU): 400mg / m2 IV bolus (15 min) followed by continuous IV infusion for 46 h of 2,400 mg / m2 on day 1 of each cycle.
  Oxaliplatin 85 mg / m2 IV over 120 minutes on cycle day 1
  Other Names: Leucovorin/Fluorouracil/Oxaliplatin
Biological: Anti-EGFR or Bevacizumab — In case of RAS wt colorectal cancer administer anti-EGFR together with FOLFOX6m, and in case of mutated RAS colorectal cancer administer Bevacizumab together with FOLFOX6m.
  Treatment administered following Summary of medicinal Product Characteristics (SmPC) approved indications.
  Other Names: monoclonal antibody anti EGFR (RASwt) or Bevacizumab (RASmut)
Drug: LIVERPEARLS-Irinotecan — Chemoembolization of Irinotecan in 100 +/- 50 micron hydrogel microspheres. Irinotecan will be loaded at a dose of 100 mg. LIFEPEARLS® is a CE marked medical device consisting of microspheres for use in chemoembolization. This device allows the continuous release of irinotecan in liver tumors causing a specific necrosis. The penetration of irinotecan into the tumor tissue is deeper thanks to the microspheres, avoiding proximal occlusion of the vessels supplying the tumor.
  Other Names: Chemoembolization of Irinotecan in hydrogel microspheres
  Arms: Experimental

SUMMARY:
Non-commercial, prospective, randomized, multicenter, national, phase II, open-label comparative clinical trial.

The patients will be randomized in a 1: 1 ratio in two arms:

Control arm. Systemic chemotherapy with FOLFOX6m + monoclonal Ab Experimental arm. Systemic chemotherapy with FOLFOX6m + monoclonal Ab + Intra-arterial liver chemotherapy with LIFEPEARLS-IRINOTECAN (catheterization and infusion of 100 +/- 50 micron microspheres loaded with 100 mg of irinotecan in both liver lobes) cycles 2 and 4.

The main objective is to evaluate the radiological objective response rate according to the RECIST version 1.1 criteria at 6 months. Secondary objectives include: Evaluate overall survival, progression-free survival (PFS), safety profile, hepatic PFS, R0 liver surgery rate.

DETAILED DESCRIPTION:
Hepatic intra-arterial therapy (TACE) with irinotecan has been used in several prospective studies demonstrating an acceptable toxicity profile. Two randomized phase II studies have evaluated the efficacy of TACE with irinotecan compared to conventional chemotherapy in metastatic colon cancer. A second-line treatment study demonstrated an increase in PFS in the TACE versus FOLFIRI treatment arm.

A prospective open, randomized, multicenter phase II study is proposed that will include patients with liver metastases of colorectal origin with poor prognostic criteria.

LIFEPEARLS® is a CE marked medical device consisting of microspheres for use in chemoembolization. The device uses 100 +/- 50 micron microspheres of hydrogel into which chemotherapeutic agents are loaded and delivered into the hepatic artery to treat liver tumors. This device allows the continuous release of irinotecan in liver tumors causing a specific necrosis. The penetration of irinotecan into the tumor tissue is deeper thanks to the microspheres, avoiding proximal occlusion of the vessels supplying the tumor.

Systemic treatment will be administered according to the usual guidelines:

-FOLFOX6m for 6 months + monoclonal Ab (cycles are repeated every 15 days) Premedication: Dexamethasone 20 mg IV + ondansetron 8mg IV

The dose of FOLFOX will be:

Leucovorin: 400 mg / m2 IV over 15 minutes on day 1 of each cycle. Fluorouracil (5-FU): 400mg / m2 IV bolus (15 min) followed by continuous IV infusion for 46 h of 2,400 mg / m2 on day 1 of each cycle.

Oxaliplatin 85 mg / m2 IV over 120 minutes on cycle day 1. In case of RAS wt colorectal cancer administer anti-EGFR together with FOLFOX6m, and in case of mutated RAS colorectal cancer administer Bevacizumab together with FOLFOX6m.

In the combination arm of systemic chemotherapy with IRINOPEARL, in the 2nd and 4th cycles, chemotherapy will be replaced by treatment with hepatic chemoembolization with IRINOPEARL.

The disease will be evaluated by CT or MRI at baseline and every 12 weeks until progression according to RECIST 1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years.
* Patients with colorectal cancer and exclusive liver metastases with poor prognostic criteria,> 3 lesions and / or size> 5 cm. Patients with a diagnosis of liver metastases with synchronous presentation or with a disease-free interval may be included. If the primary tumor has not been resected, it must be clinically stable.
* Measurable disease following RECIST version 1.1 criteria
* Adequate bone marrow function, according to:

  1. Hemoglobin ≥ 9.0 g / dl (patients with hemoglobin <9 g / dl can be transfused before inclusion in the study
  2. Platelet count ≥ 100 x 109 / L
  3. Absolute Neutrophil Count (ANC) ≥ 1.5x 109 / L
* Adequate liver function, according to:

  1. Serum bilirubin ≤ 1.5 x the upper limit of normal (ULN)
  2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x ULN.
  3. Alkaline phosphatase ≤ 5 x ULN or ≤10 x ULN in the presence of bone metastases
  4. Adequate renal function, with creatinine levels <1.5 mg / dL. Blood Ureic Nitrogen (BUN)> 50 ml / min.
  5. Albumin> 3.0 g / dL
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
* Patients capable of understanding the information and giving their written informed consent to participate in the study
* Women of childbearing potential must commit to sexual abstinence or use of barrier contraceptive methods during the study and must have a negative pregnancy test.

Exclusion Criteria:

* Extension of the disease> 50% of the liver parenchyma (evaluated by CT performed within the month prior to inclusion)
* Previous chemotherapy treatment for metastatic colorectal cancer
* Clinically significant cardiovascular diseases: cerebrovascular accident / stroke (≤ 6 months before inclusion in the trial), myocardial infarction (≤ 6 months before inclusion in the trial), unstable angina, uncontrolled hypertension, congestive heart failure of New York Heart Association (NYHA) grade II or higher or severe cardiac arrhythmia.
* History of malignancy in the last three years, except for basal cell carcinoma of the skin or carcinoma in situ of the cervix treated appropriately.
* Altered coagulation (Quick> 50%)
* Patients with active infectious processes
* Patients with any of the contraindications specified in the technical data sheet of the study drug or with allergies to some of the drugs used
* Pregnant or lactating patients
* Portal thrombosis
* Severe portal hypertension
* Extrahepatic metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Evaluated at 6 months after first investigation drug administration.
  The proportion of patients with tumor size reduction according to RECIST 1.1 criteria at 6 months

SECONDARY OUTCOMES:
Overall Survival (OS) | Through study completion, average 2 years
  Time from randomization until death from any cause. Patients still alive at the last contact or lost to follow-up will be censored.
Progression free survival | Through study completion, average 2 years. Evaluated during a total of 2 years (estimated) by CT scan or MR every 12 weeks
  Time from from the date of randomization to the date of first documented disease progression according to RECIST 1.1 criteria or the date of death due to any cause. Patients without radiological documentation of progression will be censored on the date of the last control without evidence of progression.
Frequency of adverse events | Through study completion, average 2 years
  Percentage of adverse events, laboratory alterations and treatment discontinuations observed in both treatment arms classified by type and severity (Safety)
Hepatic Progression free survival | Through study completion, average 2 years. Evaluated during a total of 2 years (estimated) by CT scan or MR every 12 weeks
  Time from from the date of randomization to the date of first documented disease progression within the liver according to RECIST 1.1 criteria or the date of death due to any cause. Patients without radiological documentation of progression will be censored on the date of the last control without evidence of progression.
Proportion of patients with liver surgery | Through study completion, average 2 years.
  Proportion of patients undergoing R0 surgery for liver metastases

CONTACTS AND LOCATIONS:
Overall Officials: Estela Pineda, M.D, Study Chair — Hospital Clinic of Barcelona; David Páez, M.D., Ph.D., Study Chair — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (8):
- Spain (8):
  - Hospital Clínic, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Parc Taulí, Sabadell, Barcelona
  - H. Univ. Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Pamplona
  - Hospital Universitari i Politècnic La Fe, Valencia, Valencia